CLINICAL TRIAL: NCT06656117
Title: Comparitive Effects of Elliptical Training vs Resistance Training on Cardiopulmonary Parameters in Post CABG Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52187 Hamna
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Bypass Graft CABG
Keywords: CABG; Elliptical training; Resistance training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: In this parallel-group randmoized control trial (RCT),post Cabag patients will br assigned to either elliptical training group or to resistance training group .This study aims to evualate the comparative effects of eliptical training vs resistance training on cardiopulmonary parameters
Who Masked: Outcomes Assessor
Masking Description: The study was single blinded,as accessor of the study were kept blind to the intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elliptical training (Experimental): * Patients in group A started with a five-minute warm-up, which included cycling on a Star Trac bike and dynamic stretching.
  * Following the warm-up, participants were instructed to perform Elliptical training after completing breathing exercises.
  * At the end of the training session, participants from both groups engaged in a five-minute gradual cool down.
  Interventions: Other: Elliptical training
- Resistance training (Experimental): * Patients in group B started with a five-minute warm-up, which included cycling on a Star Trac bike and dynamic stretching.
  * Following the warm-up, participants were instructed to perform Resistance training after completing breathing exercises.
  * At the end of the training session, participants from both groups engaged in a five-minute gradual cool down.
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Elliptical training — • Throughout the training, participants' heart rates were monitored, and they were asked to report any discomfort or unusual signs.
  Arms: Elliptical training
Other: Resistance training — • Throughout the training, participants' heart rates were monitored, and they were asked to report any discomfort or unusual signs.
  Arms: Resistance training

SUMMARY:
COMPARATIVE EFFECTS OF ELLIPTICAL TRAINING VS RESISTANCE TRAINING ON CARDIOPULMONARY PARAMETERS IN POST CABG PATIENTS

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) has been widely and increasingly used since the 1960s as a common surgical procedure to restore blood flow into the stenotic coronary arteries

. It is one of the effective ways to treat coronary artery disease, which can significantly relieve patients' myocardial ischemia and hypoxia symptoms and improve their quality of life.

Data were collected from Itefaq hospital, sehat medical complex Lahore. Borg dyspnea and quality of life (SF12) questioner were used before and after the intervention.

Assessment was done through the tool before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female age 45-55 years.
* Post Coronary Artery Bypass Grafting (CABG) patients at phase III cardiac rehabilitation were included .
* Patients who had physically active lower limbs were included .

Exclusion Criteria:

* Participants who had psychological conditions that may influence understanding or answering of questionnaire.
* Patients with other cardiac lesions combined with simultaneous surgical management, such as valvular lesions, macro vascular lesions, and ventricular wall tumors.
* Patients diagnosed with emergency CABG, minimally invasive CABG, or recurrent cardiac surgery.
* Patients with severe dysfunction of important organs such as the lung, liver, and kidney.
* Patients with recent major surgery or trauma of other parts of body.
* Pregnant or lactating women.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
modified borg dyspnea scale | 4 weeks
  The modified Borg dyspnea score is a version of the CR10; 45 it uses a scale from 0 to 10, where 0 represents no dyspnea and 10 represents maximal dyspnea. Scores are obtained at the end of the 6MWD test and reflect the maximum degree of dyspnea at any time during the walk test .
Health related quality of life(SF12) | 4 weeks
  The SF-12 Health version 2 is a generic short form health survey developed in the USA from the original SF-36. It produces two summary measures evaluating physical and mental self-perceived health; for this reason, it could be a suitable and complete tool to assess the self-perceived quality of life of university students because it allows investigating both the aspects .

CONTACTS AND LOCATIONS:
Overall Officials: Sumera Hameed, M.PHIL, Principal Investigator — Riphah International University
Locations (1):
- Sehat medical complex, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No